CLINICAL TRIAL: NCT07334379
Title: Interleukin-6 Guided Treatment With Dexamethasone or Tocilizumab in Patients Hospitalized With Acute Respiratory Symptoms - a Feasibility Study
Acronym: IDENTIFY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lorenzo delSorbo (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Lorenzo delSorbo, MD, Critical Care Medicine Department, Toronto General Hospital, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-5269; ISRCTN46157068 (Registry Identifier: ISRCTN); 296418 (Other: Health Canada)
Record Dates: First submitted 2025-11-21; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — tocilizumab; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This study is a pilot, feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Routine care only
- Tocilizumab (Experimental): Routine care + single intravenous infusion of tocilizumab at a dose of 4mg/kg of body weight (up to a max 400mg).
  Interventions: Drug: Tocilizumab (Actemra®)
- Dexamethasone (Experimental): Routine care + a 10mg of oral dexamethasone per day for up to 10 days (or until hospital discharge).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Tocilizumab (Actemra®) — Subjects randomized to the tocilizumab arm will receive a single intravenous (IV) infusion of tocilizumab, given over 1 hour. The tocilizumab will be given at a dosage of 4mg per kg of body weight, up to a maximum dose of 400 mg.
  Arms: Tocilizumab
Drug: Dexamethasone — Subjects randomized to the dexamethasone arm will receive 6 mg of dexamethasone per day, for up to 10 days, or until discharged from the hospital. Dexamethasone will be given in tablet form orally (by mouth) or through an equivalent method.
  Arms: Dexamethasone

SUMMARY:
Acute hypoxemic respiratory failure (AHRF) happens when the lungs are unable to absorb enough oxygen. The bloodstream is deprived of oxygen which can eventually lead to more severe conditions like multi-organ failure (MOF) and death. AHRF accounts for over 30% of patients to critical care units, thus novel treatments are sorely needed. Research has shown that blood levels of the inflammatory biomarker Interleukin-6 (IL-6) may be a reliable marker for predicting which patients with AHRF will progress into requiring intensive care unit (ICU) admission, MOF, and eventually death. IL-6 levels were shown to reliably peak several days before MOF, ICU admission, and death. Thus, the investigators believe that by identifying patients before the peak of their IL-6 levels, they will be able to administer early treatment to prevent the patient's condition from worsening. The aim of this study is to test the feasibility of a treatment strategy for AHRF based on IL-6 measurement in patients who are admitted to hospital care with AHRF.

Patients who are eligible for the study will have their plasma IL-6 levels measured over 2 days. Patients with elevated IL-6 levels will be randomized into 1 of 3 treatment groups: standard of care only, standard of care plus a single IV infusion of Tocilizumab, or standard of care plus treatment with oral Dexamethasone for 10 days. Patients will then be observed till discharge or up to 28 days, and a follow-up phone interview will be conducted 6 months of the end of the observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Presence of new onset of respiratory symptoms in the previous 14 days upon presentation at the emergency department. Respiratory symptoms are characterized by at least one of the following: cough, dyspnea, or requirement of oxygen supplementation
3. Requirement of inpatient hospital management

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients with known contraindications to dexamethasone or tocilizumab, or any of their components
3. Allergic reaction to tocilizumab or other monoclonal antibodies
4. Patients who are using azathioprine or cyclophosphamide
5. Active tuberculosis infection
6. Patients who have active hepatic disease or hepatic impairment
7. ALT or AST >3x upper limit of normal
8. Neutrophil count <1000/mcl
9. Platelet count <50,000/mm3
10. Hemoglobin (Hb) below 8.5 g/dL,
11. White blood cell count (WBC) below 3000/mm3
12. Absolute Neutrophil Count (ANC) below 2.0 x 109/L
13. absolute lymphocyte count below 500/mm3
14. total bilirubin above ULN
15. Triglycerides (TG) above 10 mmol/L (above 900 mg/dL)
16. Serum creatinine above 1.4 mg/dL in female patients and above 1.6 mg/dL in male patients
17. Patients already receiving systemic steroids, monoclonal antibodies or other immunosuppressive medications at the time of presentation
18. Inability to comply with the regulations to avoid conception within 28 days after enrollment
19. Admission to ICU prior to randomization
20. Immediate need for intubation
21. Imminent death
22. Clinical team refusal
23. Participation in other drug clinical trials (this criterion will be discussed with the PI)
24. Reaching >72h since hospital admission
25. Pregnancy (positive pregnancy test) or breastfeeding (which is a contraindication to tocilizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
To determine the potential recruitment rate | From enrollment to completion of the study (in including the 6-month follow-up).
To assess the proportion of eligible patients who do not have daily IL-6 measurement | Baseline (Day 0) to Day 2
To assess the proportion of eligible patients who are not randomized | Baseline (Day 0) to Day 2
To determine the rate of adherence to the assigned treatment strategy and any cross-overs | Baseline to end of 28-day observation period (or hospital discharge)
To estimate the time from hospital admission to randomization and initiation of the allocated treatment | Baseline to Day 3

SECONDARY OUTCOMES:
All cause 28-day mortality | From enrollment to completion of the 28-day observation period (or hospital discharge).
Sequential Organ Failure Assessment (SOFA) score increase of ≥2 or death | From enrollment to end of 28-day observation period (or hospital discharge).
  The SOFA (Sequential Organ Failure Assessment) scale is used to assess a patient's organ function. The SOFA score is based on 6 different systems: respiratory, cardiovascular, hepatic, coagulation, renal, and neurological. Each system is given a score from 0 (best) to 4 (worst). Total SOFA score is calculated by adding the scores for each system, with a lower total SOFA scores generally denote better overall organ function.
Development of ARDS or death | From enrollment to end of 28-day observation period (or hospital discharge).
ICU admission or death | From enrollment to end of 6-month follow-up period.
Hospital length of stay | From enrollment to end of 28-day observation period (or hospital discharge).
ICU length of stay | From enrollment to end of 28-day observation period (or hospital discharge).
Need for invasive mechanical ventilation or death | From enrollment to end of 28-day observation period (or hospital discharge).
Duration of invasive mechanical ventilation | From enrollment to end of 28-day observation period (or hospital discharge).
Health related quality of life at 6 months assessed using the 36-Item Short Form Survey (SF-36) | From enrollment to 6 months after the end of 28-day observation period (or hospital discharge)
  The SF-36 is a 36-item survey that scores patients on eight health scales: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The SF-36 is structured so higher scores on each scale generally denote a more favorable health outcome. It also includes a single item that provides an indication of perceived change in health.
Survival at 6 months | From enrollment to end of 6-month follow-up period.
Complications of steroids or tocilizumab including | From enrollment to end of 28-day observation period (or hospital discharge).
  Complications including: Hypersensitivity or allergic reaction to tocilizumab, Nosocomial infections, Neuromuscular weakness, Gastrointestinal perforations.=, Hypernatremia (serum sodium >150 mmol/L), Hyperglycemia (requiring new insulin or increased insulin dose), Hepatic dysfunction, Demyelinating disorders, Myocardial infarction or acute coronary syndrome, Malignancies, Stroke, New delirium, Neuromuscular weakness, Clinically significant gastrointestinal bleeding (requiring transfusion or endoscopy), Fetal and infant harm, and Death

OTHER OUTCOMES:
To assess reasons why eligible patients are not randomized | Baseline (Day 0) to Day 2.
  In addition to primary outcome #3: To assess the proportion of eligible patients who are not randomized, the reasons why eligible patients are not randomized will also be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada